CLINICAL TRIAL: NCT03846830
Title: INVENT VPT: Incremental Velocity Error as a New Treatment in Vestibular Rehabilitation
Brief Title: Incremental Velocity Error as a New Treatment in Vestibular Rehabilitation
Acronym: INVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Fort Belvoir Community Hospital (U.S. Federal Agency); Neuroscience Research Australia (Other); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00182654; CDMRP-PT170081 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Mild Traumatic Brain Injury; Vestibular Neuropathy
Keywords: gaze stability; balance; vestibulo-ocular reflex (VOR) gain; dizzy
MeSH Terms: conditions — Brain Concussion; Vestibular Neuronitis; Dizziness

STUDY DESIGN:
Intervention Model Description: The investigators will randomize placement in two groups of gaze stability exercises (IVE or traditional VPT). Each of the three Aims will recruit active duty service members with mTBI and dizziness from the Intrepid Spirit Center at Fort Belvoir Community Hospital (FBCH) and civilians with unilateral vestibular hypofunction from Johns Hopkins University (JHU). Inclusion criteria for the FBCH site are active duty service member with mTBI and 'vestibular' symptoms (dizziness, oscillopsia, motion sensitivity, imbalance). Inclusion criteria for the JHU site are civilians with unilateral vestibular hypofunction.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IVE/VPT 6 week Crossover (Active Comparator): Subjects will randomly be placed in one of two groups (IVE or VPT) involving daily exercise for 5 weeks, 6 weeks washout, and then crossover into the other group for a final 5 weeks. The Incremental Velocity Error (IVE) group uses a device worn on the head that delivers a moving target during head motion; while Traditional Vestibular Rehabilitation (VPT) uses the traditional eye and head turning rehabilitation exercises. Gait and balance training offered throughout each of the 5 weeks epochs of training.
  Interventions: Device: Incremental Velocity Error (IVE); Behavioral: Traditional Vestibular Rehabilitation (VPT)
- IVE/VPT 3 week Crossover (Experimental): Subjects will randomly be placed in one of two groups (IVE or VPT) involving daily exercise for 3 weeks, 3 weeks washout, and then crossover into the other group for a final 3 weeks. The Incremental Velocity Error (IVE) group uses a device worn on the head that delivers a moving target during head motion; while Traditional Vestibular Rehabilitation (VPT) uses the traditional eye and head turning rehabilitation exercises. Gait and balance training will not start until the washout period.
  Interventions: Device: Incremental Velocity Error (IVE); Behavioral: Traditional Vestibular Rehabilitation (VPT)
- IVE/VPT 3 week crossover (Active Comparator): Subjects will randomly be placed in one of two groups (IVE or VPT) involving every other day exercise for 3 weeks, 3 weeks washout, and then crossover into the other group for a final 3 weeks. The Incremental Velocity Error (IVE) group uses a device worn on the head that delivers a moving target during head motion; while Traditional Vestibular Rehabilitation (VPT) uses the traditional eye and head turning rehabilitation exercises. Gait and balance training offered throughout the 3 weeks of exercise.
  Interventions: Device: Incremental Velocity Error (IVE); Behavioral: Traditional Vestibular Rehabilitation (VPT)

INTERVENTIONS:
Device: Incremental Velocity Error (IVE) — A lightweight headband has electronics attached that detect head velocity and move a laser target at a fraction of the head velocity.
Behavioral: Traditional Vestibular Rehabilitation (VPT) — Standard of care, meta-analysis vetted, eye and head motion exercises to reduced morbidity associated with dizziness and imbalance.

SUMMARY:
The objective for this study is to compare outcome measures from vestibular rehabilitation (VPT) delivered in a traditional method against a new device Incremental Velocity Error (IVE) that improves physiologic performance of the vestibulo-ocular reflex. Participants include active duty service members with mild traumatic brain injury (mTBI) and civilians with peripheral vestibular hypofunction. The investigators will use a clinical trial cross-over design with randomization to either the control (VPT) or experimental (IVE) group and measure vestibulo-ocular reflex function as well as subjective and functional outcomes in order to investigate the best means to improve delivery of vestibular rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years old
* Service members with mTBI and civilian patients with vestibular hypofunction, both of which reports vestibular symptoms (i.e. dizziness, imbalance).

Exclusion Criteria:

* Any subjects with a self-reported history of significant ophthalmic, neuromuscular, cardiovascular (except hypertension), renal/electrolyte and psychiatric disorders
* Those with uncontrolled severe hypertension (systolic BP of >200 mm Hg and/or a diastolic BP of > 110 mmHg at rest)
* Those with a recent history of alcohol and/or drug abuse within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in vestibulo-ocular reflex (VOR) Gain | Weekly, up to 6 months
  A ratio of eye/head velocity measured using a small video camera attached to a lightweight headband. This is an off-the-shelf device commonly used in clinic. Scores typically vary between 0 and 1.2 and normal ranges are between 0.8 and 1.2.

SECONDARY OUTCOMES:
Baseline vestibular function assessed with Videonystagmography/Electronystagmography (VNG/ENG) | At first visit, up to 30 minutes.
  The VNG/ENG is a suite of tests that measure oculomotor function and vestibular function by asking subjects to follow moving targets while the eyes are recording with video (VNG) or electrodes (ENG). Also included is a warm and cold air flush into the external ear, which stimulates the 8th cranial nerve. The report includes measures of eye velocity (deg/sec), position, (deg) and acceleration (deg/sec/sec) relative to the moving targets. These data are presented in a plot that is compared to normative values provided by the company to assess baseline vestibular function.
Baseline oculomotor function assessed with Videonystagmography/Electronystagmography (VNG/ENG) | At first visit, up to 30 minutes.
  This is a standard clinical test being done to characterize baseline vestibular function.
  The VNG/ENG is a suite of tests that measure oculomotor function and vestibular function by asking subjects to follow moving targets while the eyes are recording with video (VNG) or electrodes (ENG). Also included is a warm and cold air flush into the external ear, which stimulates the 8th cranial nerve. The report includes measures of eye velocity (deg/sec), position, (deg) and acceleration (deg/sec/sec) relative to the moving targets. Data also includes velocity of eye rotations relative to healthy controls. These data are presented in a plot that is compared to normative values provided by the company to assess baseline oculomotor function.
Baseline vestibular function assessed with Vestibular Evoked Myogenic Potential (VEMP) | At first visit, up to 20 minutes.
  This is a standard clinical test being done to characterize baseline vestibular function. The VEMP test uses surface electromyography to record sternocleidomastoid and/or inferior oblique muscle activity. The report output is the latency and magnitude of the muscle response. These data are presented in a plot that is compared to normative values provided by the company to assess baseline vestibular function.
Baseline vestibular function assessed with Rotary Chair | At first visit, up to 40 minutes.
  This is a standard clinical test being done to characterize baseline vestibular function. The Rotary Chair test positions subjects in an enclosure, seated in a chair that moves 360deg at 60 and 240 deg/sec. The report includes measures of eye and head velocity (deg/sec) and position (deg). These data are presented in a plot that is compared to normative values provided by the company to assess baseline vestibular function.
Change in Dizziness Handicap Inventory | Every other week, up to 6 months
  This is a questionnaire filled out by the subject that includes items describing the behavioral impact of experiencing dizziness/imbalance. Each items is scored as a Likert scale type variable where subjects answer Yes Sometimes or No. Scores range from 0-100, with 0 indicating no impact of dizziness while scores of 100 indicate a severe impact.
Change in Activity Specific Balance Confidence scale (ABC) | Every other week, up to 6 months
  Self-report measure that asks subjects to rate their confidence performing 16 activities of daily living. Each item is scored from 0 to 100% in 10% increments with 0% indicating No confidence and 100% indicating Complete confidence.
Change in Neurobehavioral Symptom Inventory (NSI) | Every other week, up to 6 months
  This is a 22 item questionnaire that asks how bothersome symptoms are. Items are scored from 0 (None) to 4 (Very Severe). HIgher scores imply the symptoms are more bothersome.
Change in Patient Global Impression of Change (PGIC) | Every other week, up to 6 months
  This is a questionnaire filled out by the subject that assesses change in activity, symptoms, emotions, and overall quality of life. Items are between 1 (no change) to 7 (considerable) and higher scores suggest a better change in symptom management.
Change in Dynamic Visual Acuity (DVA) | Every other week, up to 6 months
  This is a standard clinical test of visual acuity during active (self-generated) head rotation. Subjects identify letters on a computer monitor; scores range from 20/10 acuity to 20/800 and normative data are available to compare.
Change in Time ( in seconds) Standing during the Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) | Every other week, up to 6 months
  Subjects stand quietly (arms folded) on the ground or on a compliant surface while time is measured up to 30 seconds. This is a standard measure of standing posture/balance. Each participant gets a score ranging from 0 to 30 seconds with higher scores correlating with a better balance.
Change in Area (in degrees) of Sway during the Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) | Every other week, up to 6 months
  Subjects stand quietly (arms folded) on the ground or on a compliant surface while sway is measured using small sensors placed on the body (inertial measurement units). The sensors measure amount of sway in degrees and the duration the subject stands is measured for up to 30 seconds. Sway scores range 0 to 20 degrees of motion side to side and fore-aft. Lower scores correlate with a better balance.
Change in the tandem walk test assessed by number of steps taken | Every other week, up to 6 months
  Ability to walk heel to toe for a distance of 10 steps.
Change in the time to complete the Timed Up and Go (TUG) Ipsi Turn. | Every other week, up to 6 months
  Subjects total time (in seconds) is recorded to stand from seated position, walk 3 meters, turn around 180-degrees and return to sit.
Change in the time to complete the Timed Up and Go (TUG) Contra Turn. | Every other week, up to 6 months
  Subjects total time (in seconds) is recorded to stand from seated position, walk 3 meters, turn around 180-degrees and return to sit.
Change in Fogginess (mental) during the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test that includes stepping while viewing a virtual scenario of a patrol task. Subjects step on/off a 6-inch step while being asked to identify objects in the virtual scene. The fogginess is rated on a visual analog scale from 0 (no symptoms) -10 (worse symptoms).
Change in Dizziness during the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test that includes stepping while viewing a virtual scenario of a patrol task. Subjects step on/off a 6-inch step while being asked to identify objects in the virtual scene. The dizziness is on a visual analog scale from from 0 (no symptoms) -10 (worse symptoms).
Change in Headache during the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test that includes stepping while viewing a virtual scenario of a patrol task. Subjects step on/off a 6-inch step while being asked to identify objects in the virtual scene. The headache is rated on a a visual analog scale from 0 (no symptoms) -10 (worse symptoms).
Change in Nausea during the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test that includes stepping while viewing a virtual scenario of a patrol task. Subjects step on/off a 6-inch step while being asked to identify objects in the virtual scene. The nausea is rated on a a visual analog scale from 0 (no symptoms) -10 (worse symptoms).
Change in visual acuity during the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test involving the use of virtual reality goggles and viewing a scenario that mimic a patrolling scenario. Subjects step on/off a 6-inch step while being asked to identify objects in the scene. A subjective rating of visual acuity using a visual analog scale from 0 (no symptoms) -10 (worse symptoms).
Change in Mean Reaction Time during the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test involve stepping on/off a 6-in step while viewing a virtual video patrol scenario. The reaction time (in milliseconds) to respond to 11 auditory cues embedded in the virtual scene is measured.
Change in 5 min heart rate during the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test involve stepping on/off a 6-in step while viewing a virtual video patrol scenario. The heart rate at 5 minute is measured in beats per minute.
Pre heart rate during the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test involve stepping on/off a 6-in step while viewing a virtual video patrol scenario. The initial heart rate is measured in beats per minute.
Post (video) heart rate during the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test involve stepping on/off a 6-in step while viewing a virtual video patrol scenario. The post video completion heart rate is measured in beats per minute.
Final heart rate during the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test involve stepping on/off a 6-in step while viewing a virtual video patrol scenario. The 3 min post video completion heart rate is measured in beats per minute.
Pre Rate of Perceived Exertion for the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test involve stepping on/off a 6-in step while viewing a virtual video patrol scenario. Rate of Perceived Exertion (RPE) is measured on a scale from 6 (rest) - 20 (maximal exertion) scale.
Post (video) Rate of Perceived Exertion for the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test involve stepping on/off a 6-in step while viewing a virtual video patrol scenario. Post RPE is measured at the end of the video using the 6 (rest) - 20 (maximal exertion) scale.
5 min Rate of Perceived Exertion for the Patrol Exertion Multitask Test (PEMT) | Every other week, up to 6 months
  This is a 12-minute test involve stepping on/off a 6-in step while viewing a virtual video patrol scenario. RPE is measured at the 5th minute from starting the video using the 6 (rest) - 20 (maximal exertion) scale.
Change in the Functional Gait Assessment (FGA) | Every other week, up to 6 months
  The FGA is a 10-item behavioral test assessing risk for fall. Each items is scored from 0 (severe) to 3 (normal) impairment. Scores range from 0 - 30 with scores compared against normative data.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Schubert, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Fort Belvoir CH, Fort Belvoir, Virginia

IPD SHARING:
Plan to Share IPD: No
We will only share de-identified individual participant data (IPD) with researchers on the approved research protocol.

REFERENCES:
- [Background] Todd CJ, Hubner PP, Hubner P, Schubert MC, Migliaccio AA. StableEyes-A Portable Vestibular Rehabilitation Device. IEEE Trans Neural Syst Rehabil Eng. 2018 Jun;26(6):1223-1232. doi: 10.1109/TNSRE.2018.2834964. PMID 29877847
- [Background] Migliaccio AA, Schubert MC. Pilot study of a new rehabilitation tool: improved unilateral short-term adaptation of the human angular vestibulo-ocular reflex. Otol Neurotol. 2014 Dec;35(10):e310-6. doi: 10.1097/MAO.0000000000000539. PMID 25122595
- [Derived] Ervin AM, Schubert MC, Migliaccio AA, Perin J, Coulibaly H, Millar JL, Roberts D, Shelhamer M, Gold D, Beauregard S, Pinto R, Brungart D, Ward BK; INVENT VPT Research Group. Incremental Velocity Error as a New Treatment in Vestibular Rehabilitation (INVENT VPT) Trial: study protocol for a randomized controlled crossover trial. Trials. 2021 Dec 11;22(1):908. doi: 10.1186/s13063-021-05876-4. PMID 34895314
- See also: Patent for the device being studied — https://www.google.com/patents/US20100198104